CLINICAL TRIAL: NCT03688230
Title: AMELION: A Randomized, Double Blinded, Phase 2, Efficacy and Safety Study of Abituzumab (EMD 525797) in Combination With Cetuximab and FOLFIRI Versus Placebo in Combination With Cetuximab and FOLFIRI in First-line RAS Wild-type, Left-sided, Metastatic Colorectal Cancer Patients With High ανβ6 Integrin Expression.
Brief Title: Study of Abituzumab in Combination With Cetuximab and FOLFIRI in Patients With Metastatic Colorectal Cancer.
Acronym: AMELION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Co-development decision
Sponsor: SFJ Pharmaceuticals X, LTD. (Industry)
Collaborators: SFJ Pharmaceuticals, Inc. (Industry); Merck KGaA, Darmstadt, Germany (Industry); AIO-Studien-gGmbH (Other); Academic and Community Cancer Research United (Other)
Responsible Party: Sponsor
Organization: SFJ Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP218797; 2018-003439-31 (EudraCT Number); AIO-KRK-0318/ass (Other: AIO-Studien-gGmbH)
Record Dates: First submitted 2018-09-24; First posted 2018-09-28 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Abituzumab; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abituzumab + Cetuximab + FOLFIRI (Experimental): Cetuximab:
  400 mg/m2 over 120 min followed by 250 mg/m2 weekly 60 min or 500 mg/m2 every two weeks, initially 120 min followed by 60 to 90 min
  * (60 min [± 5 min] after completion of the cetuximab infusion) Abituzumab 1000 mg: every 2 weeks for 60 min
  * (60 min [± 5 min] after completion of the abituzumab infusion) FOLFIRI: every 2 weeks Irinotecan 180 mg/m² IV, 30 - 90 min day 1 Folinic acid (racemic) 400 mg/m² IV, 120 min day 1 5-FU 400 mg/m² bolus day 1 5-FU 2400 mg/m² IV over a period of 46 h day 1-2
  Interventions: Drug: abituzumab
- Placebo + Cetuximab + FOLFIRI (Placebo Comparator): Cetuximab:
  400 mg/m2 over 120 min followed by 250 mg/m2 weekly 60 min or 500 mg/m2 every two weeks, initially 120 min followed by 60 to 90 min
  * (60 min [± 5 min] after completion of the cetuximab infusion) Placebo: every 2 weeks for 60 min
  * (60 min [± 5 min] after completion of the placebo infusion) FOLFIRI: every 2 weeks Irinotecan 180 mg/m² IV, 30 - 90 min day 1 Folinic acid (racemic) 400 mg/m² IV, 120 min day 1 5-FU 400 mg/m² bolus day 1 5-FU 2400 mg/m² IV over a period of 46 h day 1-2
  Interventions: Combination Product: Placebo + Cetuximab + FOLFIRI

INTERVENTIONS:
Drug: abituzumab — 1000 mg IV
  Other Names: EMD525797
  Arms: Abituzumab + Cetuximab + FOLFIRI
Combination Product: Placebo + Cetuximab + FOLFIRI — 400 mg/m2 over 120 min followed by 250 mg/m2 weekly 60 min or 500 mg/m2 every two weeks, initially 120 min followed by 60 to 90 min
  Arms: Placebo + Cetuximab + FOLFIRI

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the experimental drug abituzumab (EMD525797) in combination with cetuximab and FOLFIRI in RAS wild-type, left-sided, metastatic colorectal cancer patients with high ανβ6 integrin expression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent prior to any study specific procedure;
2. Age: ≥18 years;
3. Evidence of newly diagnosed stage IV metastatic colorectal cancer. Primary tumor location on the left side of the Colon (including left splenic flexure) or rectum;
4. Demonstrated wild-type RAS mutation status in the tumor (primary tumor or metastasis) by local assessment;
5. Tumor tissue specimen shows high ανβ6 integrin expression, as determined by central laboratory assessment;
6. Tumor tissue specimen (formalin-fixed, paraffin-embedded block) preferably from primary resection and/or if available from a surgical sample from metastatic site must be available for central laboratory based ανβ6 integrin expression analysis. (No Fine Needle Aspiration [FNA] will be accepted);
7. At least 1 radiographically documented measurable lesion in a previously non-irradiated area according to RECIST (Version 1.1), i.e., this lesion must be adequately measurable in at least 1 dimension (longest diameter to be recorded) as ≥2 cm by conventional techniques or ≥1 cm by spiral CT scan;
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
9. Females of childbearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study;

Exclusion Criteria:

1. Demonstrated any RAS or BRAF mutation;
2. Prior anti-EGFR or other targeted therapy;
3. Prior chemotherapy of the colorectal cancer, except for (neo) adjuvant therapy completed at least 6 months before randomization;
4. Radiotherapy (localized radiotherapy for pain relief is allowed to non-target lesions);
5. Investigational drug treatment for the treatment of malignancies in the past;
6. Concurrent participation in another interventional clinical study;
7. Pregnancy (exclusion confirmed with beta-hCG test) or lactation;
8. Any history or evidence of brain metastases or leptomeningeal metastases;
9. History of secondary malignancy within the past 5 years, except for basal cell carcinoma or carcinoma in situ of the cervix uteri, if treated with curative intent;
10. Concomitant chronic systemic immune or hormone therapy not indicated in this study protocol (except for physiologic replacement; steroids up to 10 mg per day of prednisone equivalent or topical and inhaled steroids are allowed);
11. Clinically relevant coronary artery disease (New York Heart Association [NYHA] functional angina classification III/IV), congestive heart failure (NYHA III/IV), or clinically relevant cardiomyopathy;
12. Uncontrolled hypertension defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg under resting conditions;
13. History of myocardial infarction in the last 12 months, or a high risk of uncontrolled arrhythmia, coagulation disorder associated with bleeding or recurrent thrombotic events, with the exception of arterial fibrillation treated with anti-coagulants;
14. Recent peptic ulcer disease (endoscopically proven) within 6 months of randomization, chronic inflammatory bowel disease, or acute/chronic ileus;
15. Active infection (requiring IV antibiotics and/or antiviral therapy), including active tuberculosis, active or chronic Hepatitis B or C, or ongoing HIV infection, AIDS;
16. Presence of any contra-indications or known hypersensitivity to treatment with abituzumab, cetuximab, and FOLFIRI, or to any of the excipients of these drugs;
17. Concomitant treatment with prohibited medications;
18. Medical or psychological conditions that would not permit the patient to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 16 months
  Progression free survival per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, as determined by investigator.

SECONDARY OUTCOMES:
Overall Survival (OS) | 68 months
  The overall survival is defined as the time from randomization to death from any cause.
Objective Response Rate (ORR) | 16 months
  ORR will be estimated as the proportion of responders in each treatment arm, defined as a patient whose best overall response is PR or better during the treatment period according to RECIST 1.1.
Depth of Response (DPR) | 16 months
  Depth of response will be estimated as the maximum percent tumor shrinkage during treatment.
Early Tumor Shrinkage (ETS) | 68 months
  ETS will be estimated as the proportion of patients achieving a ≥20 % decrease from baseline in the sum of longest tumor diameters.
Secondary Resection Rate With a Potentially Curative Intent | 16 months
  Patients for whom the resectability of metastases becomes evident during the study therapy should undergo a surgical resection of the metastases.
Number of participants with treatment-related adverse events summarized by CTCAE severity grade (v5.0). | 68 months
  Adverse events will be summarized by body system, preferred term, severity, and relationship to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Arnold, Prof. Dr., Principal Investigator — Asklepios Tumorzentrum Hamburg